CLINICAL TRIAL: NCT02641340
Title: A Phase 1, Multiple Ascending Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Fentanyl Sublingual Spray in Opioid Naive Subjects
Brief Title: Fentanyl Sublingual Spray in Opioid Naive Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INS002-15-050
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Pharmacology
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Cycle 1, Cohort 1 (Experimental): Fentanyl Sublingual Spray (FSS) low dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every four hours for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 1, Cohort 2 (Experimental): FSS low dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every two hours for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 1, Cohort 3 (Experimental): FSS low dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every hour for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 1, Cohort 4 (Experimental): FSS low dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every 30 minutes for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 2, Cohort 1 (Experimental): FSS medium dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every four hours for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 2, Cohort 2 (Experimental): FSS medium dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every two hours for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 2, Cohort 3 (Experimental): FSS medium dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every hour for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 2, Cohort 4 (Experimental): FSS medium dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every 30 minutes for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 3, Cohort 1 (Experimental): FSS high dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every four hours for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 3, Cohort 2 (Experimental): FSS high dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every two hours for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 3, Cohort 3 (Experimental): FSS high dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every hour for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV
- Cycle 3, Cohort 4 (Experimental): FSS high dose (n=6) or Fentanyl Citrate IV 50 mcg (n=2) will be administered once every 30 minutes for a maximum of three doses.
  Interventions: Drug: Fentanyl Sublingual Spray; Drug: Fentanyl Citrate IV

INTERVENTIONS:
Drug: Fentanyl Sublingual Spray — Fentanyl delivered at low, medium and high doses by sublingual spray (FSS)
  Other Names: SUBSYS®
Drug: Fentanyl Citrate IV — Fentanyl Citrate 50 mcg, delivered intravenously

SUMMARY:
The primary objective of this trial is to determine the pharmacokinetic and pharmacodynamic relationship of multiple dose administration of fentanyl sublingual spray in opioid naive participants. The secondary objective is to determine the safety and tolerability of multiple dose administration of fentanyl sublingual spray in opioid naive subjects.

DETAILED DESCRIPTION:
For all cycles, blood will be drawn according to the following schedule:

The 0 time (pre-dose) blood sample will be collected within 60 minutes prior to first study drug administration.

Cohort l: 0 (pre-dose), 5, 15 and 30 minutes after the first dose and at 1, 2, 4 (prior to second-dose), 4.083, 4.25, 4.5, 5, 6, 8 (prior to third-dose), 8.083, 8.25, 8.5, 9, 10, 12, 16 and 24 hours after the first dose.

Cohort 2: 0 (pre-dose), 5, 15 and 30 minutes after the first dose and at 1, 2 (prior to second-dose), 2.083, 2.25, 2.5, 3, 4 (prior to third-dose), 4.083, 4.25, 4.5, 5, 6, 8, 10, 12, 16 and 24 hours after the first dose.

Cohort 3: 0 (pre-dose), 5, 15, 30 and 45 minutes after the first dose and at 1 (prior to second-dose), 1.083, 1.25, l.5, 1.75, 2 (prior to third-dose), 2.083, 2.25, 2.5, 2.75, 3, 4, 8, 12, 16 and 24 hours after the first dose.

Cohort 4: 0 (pre-dose), 5, 15, 30 (prior to the second-dose), 35, and 45 minutes after the first dose and at I (prior to the third-dose), 1.083, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 4, 8, 12, 16 and 24 hours after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | within 24 hours (see detailed description)
Time to reach peak or maximum concentration following drug administration (Tmax) | within 24 hours (see detailed description)
Area under the concentration-time curve | within 24 hours (see detailed description)
  Categories: during a dosing interval (AUCtau ), from the time of dosing to infinity (AUC0-inf), from the time of dosing to the last quantifiable time point (AUC0-t)
Apparent elimination rate constant in the terminal phase by non-compartmental analysis | within 24 hours (see detailed description)
Corresponding half-life (t1/2) | within 24 hours (see detailed description)
Trough concentration during multiple dosing prior to next dose (Ctrough) | within 24 hours (see detailed description)
Accumulation ratios | within 24 hours (see detailed description)
  Categories: of Cmax (ARcmax), based on trough concentration (ARctrough), of AUCtau (ARauctau)
Dose normalized Cmax | within 24 hours (see detailed description)
Dose normalized AUC | within 24 hours (see detailed description)
  Categories: AUC0-1, AUC0-inf, AUCtau

SECONDARY OUTCOMES:
Participants with respiratory depression requiring the use of naloxone | within 24 hours
Participants with hypoxia requiring oxygen administration | within 24 hours
Participants needing noninvasive respiratory maneuvers (e.g., jaw thrust, bag-valve mask) to improve respiratory status at any point during the study | within 24 hours
Participants with hypotension requiring intervention | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc
Locations (1):
- Lotus Clinical Research, Inc., Pasadena, California, United States

REFERENCES:
- [Derived] Rauck RL, Oh DA, Singla N, Koch C, Parikh N, Nalamachu S, Yu J, James S. Pharmacokinetics of Fentanyl Sublingual Spray in Opioid-Naive Participants: Results of a Phase 1, Multiple Ascending Dose Study. Clin Drug Investig. 2018 Aug;38(8):715-726. doi: 10.1007/s40261-018-0658-9. PMID 29909433
- [Derived] Rauck RL, Oh DA, Singla N, Koch C, Parikh N, Nalamachu S, Wilson D, Yu J, Vetticaden S. Pharmacokinetics and safety of fentanyl sublingual spray and fentanyl citrate intravenous: a multiple ascending dose study in opioid-naive healthy volunteers. Curr Med Res Opin. 2017 Nov;33(11):1921-1933. doi: 10.1080/03007995.2017.1371681. Epub 2017 Sep 23. PMID 28942715